CLINICAL TRIAL: NCT01382472
Title: MICROS-Pilot Study Microcirculation In Acute Coronary Syndromes; Effect of Pre-treatment of High Dose Rosuvastatin on Coronary Microcirculation in Primary PCI
Brief Title: Microcirculation In Acute Coronary Syndromes
Acronym: MICROS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Helse Vest (Other); University Hospital of North Norway (Other); St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MICROS
Record Dates: First submitted 2011-06-20; First posted 2011-06-27 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2016-08

CONDITIONS: ST Elevation (STEMI) Myocardial Infarction
Keywords: STEMI; PPCI; Statins; Infarct size
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction | interventions — Rosuvastatin Calcium; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosuvastatin (Experimental): 40 mg rosuvastatin pre PCI and daily during hospital stay
  Interventions: Drug: Rosuvastatin
- Historical data (KOMPIS) (Other): Patients from the KOMPIS trial (n=44) will be used as historical controls. They received no statins omn the first day. Low dose simvastatin during hospital stay.
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Rosuvastatin — 40 mg per operative in PPCI, the 40 daily during hospital stay
  Other Names: Crestor-AstraZeneca
  Arms: Rosuvastatin
Drug: Simvastatin — No statin acutely. Simvastatin 20 mg from day 2.
  Arms: Historical data (KOMPIS)

SUMMARY:
In this mechanistic pilot study in 40 patients the investigators will compare the findings in patients treated with very early high dose statin therapy with historic controls from the KOMPIS study published in EHJ 200925. The investigators want to assess if early high dose statin therapy in patients treated with primary PCI:

1. reduces area of myocardial infarction, reduces volumes and improves remodelling as assessed by MRI at 2 days and at 2 months
2. improves microcirculation (Decreased number of patients with MO) as assessed by first pass time estimated with MRI 2 days
3. have impact on coronary blood flow as assessed by intravascular registrations and TIMI frame count immediately after PCI
4. reduce levels of CK-MB and TnT measured as area under the curve during the hospital stay at improves neurohumoral profile assessed by Heart Rate Variability (HRV) and neurohormones at discharge and at 2 months follow-up
5. improves endothelial function assessed by flow mediated vasodilatation at discharge
6. alters Peak VO2 at 1 and 6 month
7. reduce levels of CRP and pro-inflammatory cytokines during index hospitalization and at follow-up alters collagen turnover

DETAILED DESCRIPTION:
Impairment of the myocardial microcirculation in the setting of AMI is multifactorial in etiology. This may be due to vasoactive factors including endothelin-1, which is a potent vasoconstricting peptide and increasingly expressed in the active plaque . Oxidative stress and ischaemia per se may also reduce the bioavailability of nitric oxide, further contributing to the dysfunction of the myocardial microcirculation.

Statins have been shown to benefit ACS patients in that they are believed to decrease reperfusion injury after an ischemic event, promote plaque stabilization, and reduce inflammation in ACS patients. In patients admitted with acute coronary syndrome (ACS), treatment with statins <24 hours of presentation was associated with lower incidences of death, stroke, reinfarction, heart failure, and pulmonary edema compared with delayed administration .

40 statin naive patients admitted with STEMI will receive high dose statin Rosuvastatin 40 mg pre/per primary PCI and continue this treatment during the hospital stay. The high dose of rosuvastatin is chosen to achieve high plasma concentration as early as possible for per conditioning of the myocardium at risk. At discharge they will be switched to standard dose statin.

Myocardial infarction will be assessed with Contrast enhanced cardiac magnetic resonance at 2 days and at 2 months. Microvascular obstruction (MO) may be assessed by first- pass perfusion (FPP) and delayed hyper enhancement (DHE) MO is defined as regional hypoperfusion on first-pass perfusion as previously described . The investigators have recently demonstrated that MO as verified by CMR following MI may allow early identification of patients with a high risk of LV remodeling likely to benefit from pharmacological therapy .

Blood tests for assessment of collagen turnover, neurohumoral activation and inflammation will be drawn daily during hospital stay.

The Results will be compared with the findings of statin naive patients from tha KOMPIS trial who were not treated with high dose pre and per operative statins

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Evidence of acute ST elevation myocardial infarct.
* Planned primary PCI procedure.
* Obtained written informed consent.
* "One vessel disease"

Exclusion Criteria:

* History of previous myocardial infarction
* History of valvular disease
* Ongoing therapy for hyperlipidemia
* History of heart failure
* Any active non-cardiac co-morbidity or condition that is likely to compromise patient cooperation or survival during the follow-up period of the study.
* Pregnancy (In doubt a urine test will be employed before treatment)
* Lactating females
* Asians
* Previous muscle disease
* Reduced glomerular filtration
* Active hepatic disease
* Ongoing oral anticoagulation therapy
* Ongoing cyclosporine therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
infarct size | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alf Inge Larsen, MD, PhD, Study Chair — Helse Stavanger HF; Noreen Butt, MD, Principal Investigator — Helse Stavanger HF
Locations (3):
- Norway (3):
  - Stavanger University Hospital, Stavanger
  - University Hospital of North Norway, Tromsø
  - St. Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No